CLINICAL TRIAL: NCT01621113
Title: Restoring Lost Functions After Spinal Cord Injury: Combination Therapy With Dalfampridine and Locomotor Training for Persons With Chronic, Motor Incomplete Spinal Cord Injury
Brief Title: Combination Therapy With Dalfampridine and Locomotor Training for Chronic, Motor Incomplete Spinal Cord Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency); Acorda Therapeutics (Industry)
Responsible Party: Principal Investigator, Trevor Dyson-Hudson, M.D., Director, Spinal Cord Injury Research, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D-732-12; H133N110020 (Other Grant/Funding Number: NIDRR)
Record Dates: First submitted 2012-06-12; First posted 2012-06-18 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injuries; 4-Aminopyridine; Physical Therapy Modalities; Randomized Controlled Trial; Rehabilitation; Walking
MeSH Terms: conditions — Spinal Cord Injuries | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Locomotor Training + Dalfampridine (Experimental): Subjects randomized to this group will undergo 10 weeks of double-blind treatment with extended release dalfampridine tablets (10 mg twice daily) while simultaneously receiving locomotor training therapy (5 sessions per week x 10 weeks = 50 sessions total).
  Interventions: Drug: Dalfampridine
- Locomotor Training + Placebo (Placebo Comparator): Subjects randomized to this group will undergo identical treatment, but will take placebo tablets while simultaneously receiving locomotor training therapy (5 sessions per week x 10 weeks = 50 sessions total).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dalfampridine — Dalfampridine 10 mg tablet, twice-daily, for 10 weeks
  Other Names: Ampyra; Fampridine Sustained Release (Fampridine-SR); 4-Aminopyridine (4-AP)
  Arms: Locomotor Training + Dalfampridine
Drug: Placebo — Placebo tablet, twice daily, for 10 weeks.
  Arms: Locomotor Training + Placebo

SUMMARY:
The purpose of this study is to determine the efficacy, safety, and tolerability of treatment with dalfampridine in combination with locomotor training in persons with chronic, motor incomplete SCI.

DETAILED DESCRIPTION:
Research suggests that combining therapies could result in important gains in restoring function and improving quality of life in persons with spinal cord injury (SCI). Locomotor training is an activity-dependent rehabilitation therapy that provides repetitive stepping facilitated by manual assistance and body weight support on a treadmill. Recent studies report improvements in walking and standing in individuals with motor incomplete SCI that have undergone intensive standardized locomotor training therapy. Extended release dalfampridine (also known as fampridine or 4-aminopyridine [4-AP]) is a broad spectrum potassium channel blocker that has been shown in animal studies to increase conduction of action potentials in demyelinated axons. Dalfampridine was recently approved by the U.S. Food and Drug Administration (FDA) as a treatment to improve walking in persons with multiple sclerosis (MS). Demyelination is also a prominent feature of incomplete SCI that contributes to the clinical presentation of persons with these injuries.

The purpose of this study is to determine the efficacy, safety, and tolerability of treatment with dalfampridine in combination with locomotor training in persons with chronic, motor incomplete SCI. We hypothesize that persons undergoing combination therapy with dalfampridine and locomotor training will show significantly greater improvements in walking speed and other measures of SCI function than those receiving locomotor training alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years, inclusive;
* Neurological impairment secondary to a traumatic spinal cord injury that occurred at least twelve (12) months prior to the screening visit;
* Neurological level of the injury between C4 and T10, inclusive;
* The injury is classified as motor incomplete (AIS grade C or D);
* Able and willing to comply with the study protocol, including availability for all scheduled clinic visits and locomotor training sessions.

Exclusion Criteria:

* The participant is a lactating female, or a female of childbearing potential who is sexually active, has not had a hysterectomy or oophorectomy, and is not using an approved birth control method (e.g. tubal ligation, implantable contraception device, oral or injectable contraceptive, barrier method, or sexual activity restricted to vasectomized partner);
* The participant has a history of seizures or treatment for seizure disorders;
* The participant has renal impairment (Creatinine Clearance < 80 mL/min);
* The participant has a known allergy to pyridine-containing substances or any of the inactive ingredients of the dalfampridine;
* The participant has a clinically significant abnormal laboratory values or an abnormal electrocardiogram (ECG);
* The participant has evidence of significant, diffuse, or generalized lower motor neuron damage;
* The participant has received new concomitant medication less than 3 weeks before the study or has a dose of current concomitant medication that is expected to change during study;
* The participant has received botulinum toxin injection for spasticity within 4 months of the screening visit;
* The participant has taken any other investigational drugs within 30 days before screening;
* The participant is known to have been treated previously with dalfampridine (4 aminopyridine) in any formulation, whether through participation in a previous fampridine study or by self-medication.
* The participant has received locomotor training therapy within 6 months of the screening visit;
* The participant has a history of alcohol or drug abuse in the previous year;
* The participant has a medical condition that would interfere with interpretation of study results or study conduct.

Note: Due to equipment and safety issues associated with locomotor training, participants must weigh less than 300 lbs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-06; Primary Completion 2017-10-09 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Change in 6-Minute Walk Test (6MWT) Distance at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22) Visits
  The 6MWT measures the distance (in meters) walked within 6 minutes. The test is a measure of endurance; however, can also be used to measure walking speed.

SECONDARY OUTCOMES:
Change in 10-Meter Walk Test (10MWT) Speed at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The 10MWT measures the time in seconds that it takes a person to walk 10m. The test is a measure of functional capacity and assesses short-duration walking speed.
Change in Timed 25-foot walk (T25FW) Speed at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The T25FW is a quantitative measure of lower extremity function in persons with multiple sclerosis. The T25FW was the primary outcome measure of efficacy used in MS studies of dalfampridine and is being performed in our study as a means of comparing results across studies and populations. The T25FW can be measured during the 10MWT.
Change in Walking Index for Spinal Cord Injury II (WISCI II) Scores at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The WISCI II is a walking scale specifically developed for use in clinical trials in persons with incomplete SCI. Walking ability is scored on a 21-point ordinal scale (0-20, where 0 indicates a person is unable to stand and/or participate in assisted walking and 20 indicates a person can walk more than 10m without walking aids or physical assistance), where a lower number indicates higher impairment.
Change in Spinal Cord Injury Functional Ambulation Index (SCI-FAI) Scores at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The SCI-FAI is an observational gait assessment instrument that addresses three key domains of walking function in individuals with SCI. The three SCI-FAI subscales are Gait, Assistive Device, and Walking Mobility. Parameters of the SCI-FAI are measured during the first 2 minutes of the 6MWT (see above).
Changes on International Standards for Neurological Classification of Spinal Cord Injury at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  Neurological examination will be performed using the International Standards for Neurological Classification. Sensory scores and lower extremity motor scores are derived at the time of this exam.
Change in Lower-Extremity Motor Scores (LEMS) at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The LEMS measures strength in five muscle groups bilaterally (hip flexors, knee flexors and extensors, and ankle dorsiflexors) with the modified British Medical Research Council scale and is performed during the International Standards examination.
Change in Berg Balance Scale (BBS) Scores at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The BBS is a 14-item instrument originally designed to assess the risk for falls in community.
Change in Modified Ashworth Scale (MAS) Scores at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  Spasticity assessments will be performed at each study visit using the modified Ashworth scale (MAS). Ashworth scores will be averaged across three muscle groups bilaterally: hip adductors, knee extensors, and knee flexors. The Ashworth Scale data will be collected on a 1-5 scale rather than the published 0-4 scale.
Change in Bowel Management Questionnaire Scores at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The bowel management questionnaire uses a 6-point scale and requires the subject to rate the frequency (0, "Not at all"; 5, "Almost always") of ten items regarding bowel management over the past month.
Change in Bladder Management Questionnaire Scores at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The bladder management questionnaire uses a 6-point scale and requires the subject to rate the frequency (0, "Not at all"; 5, "Always or almost always") of eight items regarding bladder management over the past month.
Change in Female Sexual Function Index (FSFI) Scores at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The FSFI is a multidimensional, self-report instrument used to assess female sexual function. Six domains are identified that include desire, subjective arousal, lubrication, orgasm, sexual satisfaction, and pain.
Change in International Index of Erectile Function (IIEF) Scores at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The IIEF is a 15-item questionnaire to assess male sexual function. Quality of male sexual function is assessed in 5 domains, with 6 items that assess erectile function, 2 items that address orgasmic function, 2 questions that assess sexual desire, 3 items that assess intercourse satisfaction, and 2 items that assess overall sexual satisfaction.
Changes in Pulmonary Function Tests at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  Pulmonary function testing will be performed (V max Spectra 29N, Carefusion, Yorba Linda, CA) to measure spirometric parameters, static lung volumes, cough strength, and maximal mouth expiratory and inspiratory pressures.
Changes in Autonomic Function at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  To assess changes in autonomic cardiovascular function, heart rate (3 lead ECG Ivy Biomedical Systems, Inc. Branford, CT) and blood pressure (Finometer Midi, Finapres Medical Systems, Amsterdam, Netherlands) will be continuously monitored at 5 minute intervals at rest and during locomotor training.
Changes on the International Spinal Cord Injury Pain Basic Data Set (ISCIPDS:B) at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The ISCIPDS:B contains core questions about clinically relevant information concerning SCI-related pain that can be collected by health-care professionals with expertise in SCI in various clinical settings. Each person is asked to describe the three worst pain problems he/she is currently experiencing.
Change in Spinal Cord Independence Measure III (SCIM III) Scores at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The SCIM is a measure of functional ability developed specifically for individuals with SCI to evaluate their performance of activities of daily living (ADL). The SCIM III is composed of 19 items in 3 sub-scales: (a) self-care (6 items, sub-score 0-20); (b) respiration and sphincter management (4 items, sub-score 0-40); and (c) mobility (9 items, sub-score 0-40). The total score ranges from 0 to 100.
Change in Spinal Cord Injury-Functional Index (SCI-FI) Scores at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The Spinal Cord Injury Functional Index (SCI-FI) is a comprehensive, SCI-specific measure to assess functional activities related to quality of life for individuals with SCI. The SCI-FI covers five distinct functional domains: Ambulation, Basic Mobility, Fine Motor Function, Self-Care (including bowel and bladder), and Wheeled Mobility.
Change in 12-Item Short Form Health Survey (SF-12) Scores at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The SF-12 is a generic health-status measure developed by RAND to assess outcomes of medical care and has been used previously by the SCI Model Systems.
Change in Satisfaction with Life Scale (SWLS) Scores at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The SWLS is a 5-item measure of the single concept of global life satisfaction. The SWLS is currently used in the SCI Model Systems dataset and normative data for individuals with SCI is available.
Change in Craig Handicap Assessment and Reporting Technique (CHART) Scores at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The CHART is a 32-item self-report measure of major domains of participation, which has also been utilized extensively by SCI Model System researchers. It assesses functioning in 6 domains of normative role functioning: Physical Independence, Mobility, Occupation, Social Integration, Cognitive Independence, & Economic Self-Sufficiency.
Change in Subject Global Impression (SGI) of Change at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The SGI of change is a subject-rated instrument that measures change in the subject's overall status on a 7-point scale. Scores range from 1 (very much improved) to 7 (very much worse).
Change in Clinician Global Impression (CGI) of Change at 10 Weeks | Baseline, Mid-Point (Week 5), Final (Week 10), and Follow-up (Week 22)
  The study physician will rate on a 7-point scale the subject's overall clinical condition following treatment as compared to that at baseline. Scores range from 1 (very much improved) to 7 (very much worse).
Adverse Event Case Report Form | Every two weeks for 10 weeks
  Adverse experience(s) will be recorded on the Adverse Event Case Report Form, including the date and time of onset, severity, the relationship to study intervention, the date of resolution, the action taken, and the outcome of the adverse experience. The responsible physician will make a causality assessment for every adverse experience.
Side Effects Record | Every two weeks for 10 weeks
  Participants will be provided a list of side-effects associated with dalfampridine treatment. Three lines marked "other" for open-choice responses will accompany the selection of options for forced-choice side-effects. Participants will rate the severity (visual analog scale [VAS]; 0-100) and frequency ("never", "occasionally", "sometimes", "often" or "always") of side effects for each of the forced and open choice answers. Severity and frequency of side-effects will be rated by participants every 2 weeks during the intervention part of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Steven C. Kirshblum, M.D., Principal Investigator — Kessler Institute for Rehabilitation; Gail F. Forrest, Ph.D., Principal Investigator — Kessler Foundation; Trevor A. Dyson-Hudson, M.D., Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Institute for Rehabilitation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided